CLINICAL TRIAL: NCT02594969
Title: The Effect of Diluted Sodium Hypochlorite Solution and Moisturizers on Skin Barrier Function in Atopic Dermatitis
Acronym: AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 523979
Record Dates: First submitted 2014-07-10; First posted 2015-11-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Group (Active Comparator): These subjects do not have atopic dermatitis and are considered healthy. They will participate in the bleach bath and the moisturizer application.
  Interventions: Other: Bleach Bath and Moisturizers
- Atopic Dermatitis Group (Experimental): These subjects have atopic dermatitis and are considered healthy. They will participate in the bleach bath and the moisturizer application.
  Interventions: Other: Bleach Bath and Moisturizers

INTERVENTIONS:
Other: Bleach Bath and Moisturizers — All subjects will have one forearm in a bleach bath and the other forearm in a water bath for 10 minutes. Following the bath, skin barrier function will be evaluated. Secondly, moisturizers will be applied to the arms and the skin barrier will be evaluated overtime.
  Other Names: Hypochlorite Solution

SUMMARY:
The goal is this study is to investigate the effects of dilute bleach on the skin of subjects with atopic dermatitis and those with healthy skin. The second goal is to evaluate the effects of different moisturizers on the skin barrier of subjects with and without atopic dermatitis. The investigators hypothesize that the bleach bath will increase the skin pH, decrease the skin hydration, and increase skin water loss in all study subjects. Secondly, the investigators hypothesize that moisturizers with the lowest pH and the highest water to oil ratio will result in improved skin barrier function. Furthermore, the investigators believe there will be a greater improvement in patients with atopic dermatitis.

DETAILED DESCRIPTION:
The study has two main parts. Subjects in both groups will have one forearm in a dilute bleach bath and the other arm in a water bath for 10 minutes. The change in skin will be measured using different painless devices. The second part of the study involves application of 4 various moisturizers. The change in skin will be measured over a period of time using the non-invasive devices.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 years to 65 years
* Has been diagnosed with atopic dermatitis by a board-certified dermatologist at UC Davis
* Subject/parents/legal guardians able to read and comprehend the study procedure and consent forms.

Exclusion Criteria:

* Those who are pregnant, prisoners, or cognitively impaired
* Those who do not fit the inclusion criteria

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in transepidermal water loss post-bath immersion | 10 minutes post-bath immersion
  Subjects will immerse one randomized arm in a bleach bath and the other arm in a water bath for 10 minutes. The skin barrier function will be evaluated for change in transepidermal water loss after 10 minutes of bath immersion.

SECONDARY OUTCOMES:
Change in transepidermal water loss after moisturizer application | up to 60 minutes post-moisturizer application
  Each subject will have 4 various moisturizers placed on each arm. The skin barrier function will be measured for change in transepidermal water loss to 60 minutes post-application..
Change in skin hydration after moisturizer application | up to 60 minutes post-moisturizer application
  Each subject will have 4 various moisturizers placed on each arm. The skin barrier function will be measured for change in skin hydration up to 60 minutes post-application..
Change in skin pH after moisturizer application | up to 60 minutes post-moisturizer application
  Each subject will have 4 various moisturizers placed on each arm. The skin barrier function will be measured for change in skin pH up to 60 minutes post-application..
Change in skin hydration post-bath immersion | 10 minutes post-bath immersion
  Subjects will immerse one randomized arm in a bleach bath and the other arm in a water bath for 10 minutes. The skin barrier function will be evaluated for change in skin hydration after 10 minutes of bath immersion.
Change in skin pH post-bath immersion | 10 minutes post-bath immersion
  Subjects will immerse one randomized arm in a bleach bath and the other arm in a water bath for 10 minutes. The skin barrier function will be evaluated for change in skin pH after 10 minutes of bath immersion.

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- [Background] Eichenfield LF. Consensus guidelines in diagnosis and treatment of atopic dermatitis. Allergy. 2004 Aug;59 Suppl 78:86-92. doi: 10.1111/j.1398-9995.2004.00569.x. PMID 15245365
- [Background] Hanifin JM, Cooper KD, Ho VC, Kang S, Krafchik BR, Margolis DJ, Schachner LA, Sidbury R, Whitmore SE, Sieck CK, Van Voorhees AS. Guidelines of care for atopic dermatitis, developed in accordance with the American Academy of Dermatology (AAD)/American Academy of Dermatology Association "Administrative Regulations for Evidence-Based Clinical Practice Guidelines". J Am Acad Dermatol. 2004 Mar;50(3):391-404. doi: 10.1016/j.jaad.2003.08.003. No abstract available. PMID 14988682
- [Background] Rippke F, Schreiner V, Doering T, Maibach HI. Stratum corneum pH in atopic dermatitis: impact on skin barrier function and colonization with Staphylococcus Aureus. Am J Clin Dermatol. 2004;5(4):217-23. doi: 10.2165/00128071-200405040-00002. PMID 15301569
- [Background] Ryan C, Shaw RE, Cockerell CJ, Hand S, Ghali FE. Novel sodium hypochlorite cleanser shows clinical response and excellent acceptability in the treatment of atopic dermatitis. Pediatr Dermatol. 2013 May-Jun;30(3):308-15. doi: 10.1111/pde.12150. PMID 23617366
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical